CLINICAL TRIAL: NCT00469755
Title: A Comparison of Differin® Gel, 0.1% vs. Tazorac® Cream, 0.1% vs. Differin® Gel, 0.1% 6-week Treatment Switched to Tazorac® Cream, 0.1% 6-week Treatment in Patients With Acne Vulgaris
Brief Title: Differin® Gel x12 Wks vs Tazorac® Cream x12 Wks vs Differin® x6 Wks Switched to Tazorac® x6 Wks for Treatment of Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Ronald W. Gottschalk, MD / Medical Director, Galderma Laboratories, L.P.
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: US10026
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2008-03

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Differin® Gel, 0.1% for 12 weeks
  Interventions: Drug: Adapalene Gel, 0.1%
- 2 (Active Comparator): Tazorac® Cream, 0.1% for 12 weeks
  Interventions: Drug: Tazarotene Cream, 0.1%
- 3 (Active Comparator): Differin® Gel, 0.1% for 6 weeks switched to Tazorac® Cream, 0.1% for 6 weeks
  Interventions: Drug: Adapalene Gel, 0.1% + Tazarotene Cream, 0.1%

INTERVENTIONS:
Drug: Adapalene Gel, 0.1% — Apply once daily in the evening for 12 weeks
  Other Names: Differin® Gel, 0.1%
  Arms: 1
Drug: Tazarotene Cream, 0.1% — Apply once daily in the evening for 12 weeks
  Other Names: Tazorac® Cream, 0.1%
  Arms: 2
Drug: Adapalene Gel, 0.1% + Tazarotene Cream, 0.1% — Apply adapalene Gel, 0.1% once daily in the evening for 6 weeks and Tazarotene Cream, 0.1% once daily in the evening for 6 weeks
  Other Names: Differin® Gel, 0.1% and Tazorac® Cream, 0.1%
  Arms: 3

SUMMARY:
To determine the efficacy and safety of 12 weeks of treatment with Differin Gel, 0.1% compared to 12 weeks of treatment with Tazorac Cream, 0.1% and compared to 6 weeks treatment with Differin Gel, 0.1% followed by 6 weeks of treatment with Tazorac Cream

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a minimum of 20 inflammatory lesions (papules and pustules) on the face
* Subjects with a minimum of 15 and a maximum of 100 non-inflammatory lesions (open comedones and closed comedones) on the face, excluding the nose

Exclusion Criteria:

* Subjects with more than 3 nodulo-cystic lesions

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 302 (Actual)
Dates: Start 2006-02; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Efficacy - total lesion counts | 12 weeks

SECONDARY OUTCOMES:
Safety - tolerability assessments and adverse event reporting | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (12):
- United States (12):
  - Therapeutics Clinical Research, San Diego, California
  - Henry Ford Medical Center-Dept. of Dermatology, Detroit, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - State University of New York Downstate Medical Center-Dept. of Dermatology, Brooklyn, New York
  - Dermatology Research Associates, Cincinnati, Ohio
  - Phoebe Rich, MD & Associates, Portland, Oregon
  - Milton S. Hershey Medical Center Center-Div. of Dermatology, Hershey, Pennsylvania
  - DermResearch, Inc., Austin, Texas
  - J & S Studies, Inc., Bryan, Texas
  - Stephens & Associates, Carrollton, Texas
  - Dermatology Research Center, Salt Lake City, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia